CLINICAL TRIAL: NCT07121036
Title: Phase I Clinical Study of a New High - Dose Vitamin C Infusion Regimen Based on Pharmacokinetic Characteristics in Combination With Standard Systemic Therapy for Patients With Advanced Malignant Solid Tumors
Brief Title: High - Dose Vitamin C Infusion Regimen Based on Pharmacokinetic Characteristics for Patients With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Professor and Doctor of Zhongnan Hospital, Zhongnan Hospital
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDVC-01
Record Dates: First submitted 2025-07-15; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Vitamin C
Keywords: High - dose Vitamin C; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single - center, multi - arm, open - label, Phase I clinical study. Referring to the progress of domestic and foreign clinical studies, 3 different high - dose vitamin C intravenous drip regimens are designed. It is planned to enroll 18 patients (6 patients in each group) with advanced malignant solid tumors. All patients will receive standard systemic anti - tumor therapy (including chemotherapy, targeted therapy, and immunotherapy). High - dose vitamin C intravenous drip treatment in different regimens will be combined on the basis of standard anti - tumor systemic therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): HDVC is intravenously dripped at a dose of 0.5 g/kg once a day
  Interventions: Drug: high - dose vitamin C
- Arm 2 (Experimental): HDVC is intravenously dripped at a dose of 0.5 g/kg twice a day
  Interventions: Drug: high - dose vitamin C
- Arm 3 (Experimental): HDVC is intravenously dripped at a dose of 0.75 g/kg twice a day
  Interventions: Drug: high - dose vitamin C

INTERVENTIONS:
Drug: high - dose vitamin C — Different dose of high - dose vitamin C in arm1, 2 and 3

SUMMARY:
Vitamin C is an essential water - soluble vitamin for the human body. It plays an important role in various physiological processes as an antioxidant and cofactor for multiple enzymes. Most vertebrates can synthesize vitamin C by themselves, but humans can only obtain it from the diet due to inactivating mutations in the synthesis enzyme gene. The incidence of severe malnutrition in tumor patients is 58.2%, and they often have insufficient intake. Vitamin C can be used for the prevention and treatment of various diseases, including vitamin C deficiency, iron - deficiency anemia, atherosclerosis, and COVID - 19. Its role in anti - tumor treatment was first proposed by Cameron E and Pauling LN in the 1970s. However, it was not verified in a subsequent randomized controlled study at the Mayo Clinic, and this treatment has been controversial ever since. Until subsequent studies found that this difference may be due to different administration routes. Oral administration is limited by absorption, transportation, and metabolism. Even at the maximum tolerated dose, the plasma drug concentration is always < 250 μmol/L, while intravenous injection can safely reach a pharmacological plasma concentration of 25 - 30 mmol/L, which is the key to exerting the anti - tumor effect. Therefore, intravenous injection of high - dose vitamin C (HDVC) as an emerging anti - tumor therapy has received renewed attention. A series of clinical studies have confirmed that a dose of 75 - 100 g/day (1.5 - 2.2 g/kg) is safe. Most pre - clinical experiments suggest that HDVC can inhibit the development or metastasis of tumors, significantly improve the survival rate of experimental animals, and prolong their survival time. It also has a synergistic or sensitizing effect on chemotherapy, radiotherapy, and targeted therapy. However, the number of clinical trials with positive results is very limited. Only a small number of studies have reported trends of increased disease control and objective response rates. For example, when combined with gemcitabine in the treatment of pancreatic cancer, the overall survival (OS) and progression - free survival (PFS) of patients were prolonged (21.7 months vs. 11.1 months; 13.7 months vs. 4.6 months). Currently, all clinical trials lack standardization and normativity in efficacy detection, and the repeatability of the experiments is poor. This has led to a situation where pre - clinical research shows good results, but clinical translation is very difficult. This may be closely related to the pharmacokinetic characteristics of vitamin C: a short half - life of only 30 minutes, high lability, first - order kinetic elimination, and rapid excretion through the kidneys. It is easily metabolized by the body's antioxidant system (especially reduced glutathione). After the infusion stops, the plasma vitamin C concentration drops rapidly, resulting in insufficient duration of the drug peak concentration or effective concentration to kill tumor cells in the body. Therefore, ensuring sufficient blood drug concentration, prolonging the duration of the effective concentration, and inhibiting the metabolism of antioxidants may improve the therapeutic effect of HDVC. This study attempts to summarize the clinical synergistic strategies of HDVC from existing clinical trials and explore a better HDVC treatment regimen. Based on comprehensive clinical research, we take patients with advanced malignant solid tumors receiving systemic anti - tumor treatment as the research objects. While patients are undergoing systemic anti - tumor treatment, HDVC treatment is combined. Three cohorts are designed: 0.5 g/kg once a day; 0.5 g/kg twice a day; 0.75 g/kg twice a day. All are intravenously dripped continuously for 5 - 7 days during the first cycle of standard systemic anti - tumor therapy, and the blood concentration of vitamin C is detected daily. The main objectives of this study are to study the pharmacokinetic characteristics of different high - dose vitamin C intravenous drip regimens in patients with advanced solid tumors, evaluate whether twice - daily administration can increase the blood concentration of vitamin C, and explore the appropriate regimen for combining high - dose vitamin C intravenous drip with standard systemic therapy in treating patients with advanced malignant solid tumors, providing ideas and a basis for the standardized clinical application of HDVC in the future.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 - 75 years old, regardless of gender. 2. The subject voluntarily participates, gives full informed consent, signs a written informed consent form, and has good compliance.

  3. Histologically or cytologically pathologically diagnosed as advanced or metastatic malignant solid tumor.

  4. Physical function status: Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.

  5. The patient must have at least one measurable lesion (RECIST 1.1). 6. Sufficient bone marrow, liver, kidney, and heart function were recorded within 7 days before enrollment, and the patient is suitable for routine chemotherapy indicated clinically according to normal care standards.

  7. No history of calcium oxalate kidney stones. 8. Expected survival ≥ 12 weeks. 9. Pathological immunohistochemistry requires a negative catalase result. 10. Patients who are undergoing systemic anti - tumor treatment and have disease progression can also enter the protocol, continue the same treatment or start a different chemotherapy regimen without interruption.

Exclusion Criteria:

* 1. Lack of pathological diagnosis of malignant solid tumor. 2. The patient currently has central nervous system (CNS) metastasis or a history of brain metastasis.

  3. Severe gastrointestinal diseases, including active bleeding. 4. Patients with severe or uncontrolled infections, heart or nervous system diseases.

  5. Major surgery within 4 weeks or local radiotherapy within 7 days before the administration of the study drug.

  6. Dementia or severe mental status changes that prevent obtaining informed consent.

  7. Women of childbearing potential must use an acceptable contraceptive method during the study and must undergo a pregnancy test within 7 days after the first chemotherapy.

  8. The patient currently has poorly controlled diabetes (fasting blood glucose (FBG) > 10 mmol/L).

  9. Glucose - 6 - phosphate dehydrogenase (G6PD) deficiency or hereditary spherocytosis.

  10. Active pulmonary tuberculosis (TB), patients who are undergoing anti - tuberculosis treatment or have received anti - tuberculosis treatment within 1 year before the first drug administration; patients with positive human immunodeficiency virus (HIV) antibodies; or patients with syphilis infection.

  11. Active viral hepatitis. If HBsAg (+) and/or HBcAb (+), HBV DNA must be < 500 IU/mL, and during the study, the patient must continue the original anti - HBV treatment throughout the process or start using entecavir or tenofovir throughout the process. Patients with positive hepatitis C virus (HCV) ribonucleic acid (RNA) must receive antiviral treatment according to local standard treatment guidelines and have liver function within Grade 1 elevation of NCI - CTCAE Version 5.0.

  12. Any abnormal laboratory values or medical conditions that, in the judgment of the investigator, make the patient unfit for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetic characteristics | from baseline to day 7
  Detect the change in vitamin C blood concentration levels from baseline to day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China